CLINICAL TRIAL: NCT01038193
Title: Cognitive Dysfunction After Aneurysmal Subarachnoid Haemorrhage
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, George KC Wong, Professor (Clinical), Chinese University of Hong Kong
Other Study IDs: GW004
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Cognitive Dysfunction
Keywords: Cognition, subarachnoid hemorrhage.
MeSH Terms: conditions — Cognitive Dysfunction; Subarachnoid Hemorrhage | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- aSAH patients: Cognitive assessment
  Interventions: Other: Cognitive assessment

INTERVENTIONS:
Other: Cognitive assessment — Cognitive and functional assessments at 2-4 weeks, 3 months and 12 months.
  Other Names: Cognition

SUMMARY:
This is a longitudinal, multi-center, prospective study of aneurysmal subarachnoid haemorrhage patients in neurosurgical units in Hong Kong.

DETAILED DESCRIPTION:
The investigators aim to recruit a total of 240 aneurysmal subarachnoid haemorrhage patients. The schedule for neuropsychological and functional assessments will be phased in at the second to third week, the third month, and the twelve months after the initial haemorrhage.

ELIGIBILITY:
Inclusion criteria

1. Spontaneous subarachnoid haemorrhage with intracranial aneurysms as aetiology
2. Admission within 96 hours of ictus
3. Aged between 21 and 75 years
4. A speaker of Chinese (Mandarin or Cantonese)
5. Informed consent from patients or their legally acceptable representatives

Exclusion criteria

1. History of previous cerebrovascular disease or neurological disease other than intracranial aneurysm
2. History of neurosurgical operation prior to ictus

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Aneurysmal subarachnoid hemorrhage patients
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2009-03-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Cognitive dysfunction | 3 and 12 months
  Montreal Cognitive Assessment

SECONDARY OUTCOMES:
Neurological Outcome | 3 and 12 months
  Modified Rankin Scale
Generic Quality of Life | 3 and 12 months
  ShortForm36(SF-36)
Activity of Daily Living | 3 and 12 months
  Barthel Index
Disease-specific Quality of Life | 3 and 12 months
  Stroke-specific-QOL
Functional Outcome | 3 and 12 months
  Functional Independent Measure (FIM)

CONTACTS AND LOCATIONS:
Overall Officials: George KC Wong, Principal Investigator — Division of Neurosurgery, CUHK
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong GK, Lam SW, Wong A, Ngai K, Mok V, Poon WS. Early Cognitive Domain Deficits in Patients with Aneurysmal Subarachnoid Hemorrhage Correlate with Functional Status. Acta Neurochir Suppl. 2016;122:129-32. doi: 10.1007/978-3-319-22533-3_26. PMID 27165892
- [Derived] Wong GK, Wong A, Zee BC, Poon WS, Chan MT, Gin T, Siu DY, Mok VC. Cognitive outcome in acute simvastatin treatment for aneurysmal subarachnoid hemorrhage: A propensity matched analysis. J Neurol Sci. 2015 Nov 15;358(1-2):58-61. doi: 10.1016/j.jns.2015.08.013. Epub 2015 Aug 12. PMID 26285662
- [Derived] Chu AC, Wong GK, Lam SW, Wong A, Ngai K, Poon WS, Mok V. Cognitive impairment in aneurysmal subarachnoid hemorrhage patients with delayed cerebral infarction: prevalence and pattern. Acta Neurochir Suppl. 2015;120:303-6. doi: 10.1007/978-3-319-04981-6_51. PMID 25366641
- [Derived] Wong GK, Lam SW, Wong A, Lai M, Siu D, Poon WS, Mok V. MoCA-assessed cognitive function and excellent outcome after aneurysmal subarachnoid hemorrhage at 1 year. Eur J Neurol. 2014 May;21(5):725-30. doi: 10.1111/ene.12363. Epub 2014 Jan 28. PMID 24471651
- [Derived] Wong GK, Lam SW, Wong A, Mok V, Siu D, Ngai K, Poon WS. Early MoCA-assessed cognitive impairment after aneurysmal subarachnoid hemorrhage and relationship to 1-year functional outcome. Transl Stroke Res. 2014 Apr;5(2):286-91. doi: 10.1007/s12975-013-0284-z. Epub 2013 Sep 7. PMID 24323708
- [Derived] Wong GK, Lam SW, Ngai K, Wong A, Poon WS, Mok V. Development of a short form of Stroke-Specific Quality of Life Scale for patients after aneurysmal subarachnoid hemorrhage. J Neurol Sci. 2013 Dec 15;335(1-2):204-9. doi: 10.1016/j.jns.2013.09.033. Epub 2013 Oct 2. PMID 24120271
- [Derived] Wong GK, Lam SW, Ngai K, Wong A, Siu D, Poon WS, Mok V; Cognitive Dysfunction after Aneurysmal Subarachnoid Hemorrhage Investigators. Cognitive domain deficits in patients with aneurysmal subarachnoid haemorrhage at 1 year. J Neurol Neurosurg Psychiatry. 2013 Sep;84(9):1054-8. doi: 10.1136/jnnp-2012-304517. Epub 2013 Apr 20. PMID 23606736
- [Derived] Wong GK, Lam SW, Wong A, Ngai K, Poon WS, Mok V. Comparison of montreal cognitive assessment and mini-mental state examination in evaluating cognitive domain deficit following aneurysmal subarachnoid haemorrhage. PLoS One. 2013;8(4):e59946. doi: 10.1371/journal.pone.0059946. Epub 2013 Apr 3. PMID 23573223
- [Derived] Wong GK, Lam S, Ngai K, Wong A, Mok V, Poon WS; Cognitive Dysfunction after Aneurysmal Subarachnoid Haemorrhage Investigators. Evaluation of cognitive impairment by the Montreal cognitive assessment in patients with aneurysmal subarachnoid haemorrhage: prevalence, risk factors and correlations with 3 month outcomes. J Neurol Neurosurg Psychiatry. 2012 Nov;83(11):1112-7. doi: 10.1136/jnnp-2012-302217. Epub 2012 Jul 31. PMID 22851612